CLINICAL TRIAL: NCT00101725
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of TRN 002 (Crofelemer) for the Symptomatic Treatment of Diarrhea-Predominant Irritable Bowel Syndrome (d-IBS)
Brief Title: A Study of Crofelemer to Treat Diarrhea Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Michelle Widmann, Salix Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRN 002 201
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Irritable Bowel Syndrome; Colonic Diseases; Diarrhea; Gastrointestinal Disease
Keywords: Diarrhea; IBS; Irritable Bowel Syndrome; Abdominal pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Colonic Diseases; Diarrhea; Gastrointestinal Diseases; Abdominal Pain | interventions — crofelemer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 125 mg crofelemer (Experimental)
  Interventions: Drug: crofelemer
- 250 mg crofelemer (Experimental)
  Interventions: Drug: crofelemer
- 500 mg crofelemer (Experimental)
  Interventions: Drug: crofelemer
- placebo (Placebo Comparator)
  Interventions: Drug: crofelemer

INTERVENTIONS:
Drug: crofelemer

SUMMARY:
This study is designed to evaluate the safety and effectiveness of an investigational drug, TRN-002 (crofelemer) to relieve the symptoms of diarrhea-predominant irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
The investigational drug is a natural product taken from a plant that grows in South America. The study medication will be administered orally twice a day. Subjects who are eligible to participate will have a 75% chance of receiving TRN-002 and a 25% chance of receiving placebo (a substance that looks similar to TRN 002 but has no activity). Subjects will not be able to remain on certain standard IBS medications (antidiarrheals) while participating in the study. The total duration is 16 weeks.

The study requires five study visits that include physical exams, ECG and blood draws for laboratory studies. A colon procedure (such as a colonoscopy or flexible sigmoidoscopy) may also be required if it has not been performed since your diagnosis and within the last 5 years. Participants will be asked to make daily entries into a touch-tone telephone diary on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diarrhea predominant Irritable Bowel Syndrome
* Willingness to make daily calls on a touch-tone telephone
* Willingness to have an endoscopic and/or radiologic bowel evaluation, if you have not received one since your IBS diagnosis and in the past 5 years
* Willingness to use an approved method of birth control

Exclusion Criteria:

* Serious medical or surgical conditions
* Gastrointestinal Cancers, Crohns Disease or Ulcerative Colitis
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2004-12; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety of TRN-002 when administered twice daily for 12 consecutive weeks.

SECONDARY OUTCOMES:
To assess the efficacy of TRN-002 when administered twice daily for 12 consecutive weeks.

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Clinical Research Associates, Huntsville, Alabama
  - Radiant Research Phoenix Southeast, Chandler, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - AGMG Clinical Research Institute, Anaheim, California
  - Community Clinical Trials, Orange, California
  - AGMG Clinical Research, Orange, California
  - Institute of Healthcare Assessment, Inc., San Diego, California
  - Washington Gastroenterology, Washington D.C., District of Columbia
  - Consultants for Clinical Research of South Florida, Boynton Beach, Florida
  - University Clinical Research DeLand, DeLand, Florida
  - nTouch Research, Peoria, Illinois
  - Synergy Medical Education Alliance, Saginaw, Michigan
  - CRC of Jakson, Jackson, Mississippi
  - Mercy Medical Group, St Louis, Missouri
  - Tobey Village Office Park, Pittsford, New York
  - LeBauer Research Associates, PA, Greensboro, North Carolina
  - Medoff Medical / Vital Research, Greensboro, North Carolina
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - Piedmont Medical Research Assoc., Inc., Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Radient Research, Columbus, Ohio
  - Grandview Medical Research, Inc, Sellersville, Pennsylvania
  - Anderson Gastroenterology, Anderson, South Carolina
  - TriCities Medical Research, Bristol, Tennessee
  - ClinSearch, Chattanooga, Tennessee
  - Jackson Clinic, Jackson, Tennessee
  - Memphis Gastroenterology, Memphis, Tennessee
  - Radiant Research Dallas-North, Dallas, Texas
  - Tacoma Digestive Disease Research Center, Tacoma, Washington